CLINICAL TRIAL: NCT01160718
Title: Fulvestrant With or Without AZD6244, a Mitogen-Activated Protein Kinase Kinase (MEK) ½ Inhibitor, in Advanced Stage Breast Cancer Progressing After Aromatase Inhibitor: A Randomized Placebo-Controlled Double-Blind Phase II Trial
Brief Title: Fulvestrant With or Without AZD6244 in Treating Patients With Advanced Breast Cancer That Progressed After Aromatase Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAKK 21/08; SWS-SAKK-21/08; EUDRACT-2010-019965-27; EU-21046; CDR0000680800
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-positive breast cancer; HER2-positive breast cancer; HER2-negative breast cancer; progesterone receptor-positive breast cancer; recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; AZD 6244

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Fulvestrant / AZD6244 (Active Comparator): Fulvestrant 500mg i.m. day 1, 15, day 1 of cycle 2, then every 28 +/- 3 days AZD6244 75 mg p.o. bid
  Interventions: Drug: fulvestrant; Drug: selumetinib
- Arm B: Fulvestrant / Placebo (Placebo Comparator): Fulvestrant 500mg i.m. day 1, 15, day 1 of cycle 2, then every 28 +/- 3 days Placebo 3 caps p.o. bid (same appearance as AZD6244)
  Interventions: Drug: fulvestrant

INTERVENTIONS:
Drug: fulvestrant — Arm A: Fulvestrant 500mg i.m. day 1, 15, day 1 of cycle 2, then every 28 +/- 3 days Arm B: Fulvestrant 500mg i.m. day 1, 15, day 1 of cycle 2, then every 28 +/- 3 days
  Other Names: ZD9238
Drug: selumetinib — AZD6244 75 mg p.o. bid
  Other Names: AZD6244
  Arms: Arm A: Fulvestrant / AZD6244

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using fulvestrant may fight breast cancer by blocking the use of estrogen by the tumor cells. AZD6244 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether fulvestrant is more effective with or without AZD6244 in treating patients with advanced breast cancer.

PURPOSE: This randomized phase II trial is studying how well fulvestrant works with or without AZD6244 in treating patients with advanced breast cancer that progressed after aromatase inhibitor therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the efficacy of fulvestrant with versus without MEK inhibitor AZD6244 in patients with advanced stage, endocrine-sensitive breast cancer that progressed after aromatase inhibitor therapy.

Secondary

* To assess the safety and tolerability of this regimen in these patients.
* To examine other outcome parameters.
* To develop a virtual tissue bank for future translational research.

OUTLINE: This is a multicenter study. Patients are stratified according to center, prior treatment with tamoxifen citrate (yes vs no), the setting in which prior aromatase inhibitor was given (adjuvant treatment vs advanced stage treatment), HER-2 disease (positive vs negative), visceral metastasis (present vs absent), performance status (0 vs 1 or 2), and disease (measurable disease vs bone-only disease or small but unequivocal liver or lung metastases). Patients are randomized to 1 of 2 treatment arms.

* Arm I (experimental): Patients receive fulvestrant intramuscularly (IM) on days 1 and 15 of course 1 and on day 1 of each subsequent course. Patients also receive oral AZD6244 twice daily on days 1-28. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (control): Patients receive fulvestrant as in arm I. Patients also receive oral placebo twice daily on days 1-28. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Not amenable to curative therapy
* HER-2 positive disease allowed
* Disease relapse or progression after aromatase inhibitor as adjuvant therapy or for advanced stage disease
* Bilateral breast cancer allowed provided tumor endocrine sensitivity has been proven on both sides
* Measurable disease according to RECIST criteria v1.1 or other lesions assessable by radiological exams (i.e., bone-only disease or small but unequivocal liver or lung metastases)
* Received no more than 1 line of chemotherapy for advanced stage disease
* Estrogen receptor- and/or progesterone receptor-positive (≥ 10% tumor cells positive by immunohistochemistry or ≥ 10 fmol/mg cytosol protein by ligand binding assay)
* No known CNS metastases

  * Patients with brain metastases treated with radiotherapy and without any sign of brain progression after ≥ 3 months since the end of radiotherapy may be considered eligible after trial chair approval)

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Postmenopausal
* Hemoglobin ≥ 90 g/L
* Platelet count ≥ 100 x 10^9/L
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Creatinine clearance ≥ 30 mL/min
* ALT ≤ 2.5 times upper limit of normal (ULN) (≤ 5 times ULN in patients with liver metastases)
* Bilirubin ≤ 1.5 times ULN
* INR < 1.6
* PTT normal
* LVEF ≥ 50%
* Able to swallow AZD6244/placebo capsules
* Capable of understanding information given by the investigator on the trial
* Must adhere to and be geographically proximal to allow for proper staging, treatment, and follow up
* No contraindication for intramuscular injections
* No bleeding diathesis
* No current or prior malignancy other than breast cancer within the past 5 years, except carcinoma in situ of the cervix or basal cell carcinoma of the skin treated curatively
* No serious underlying medical condition that, in the judgment of the investigator, would impair the ability of the patient to participate in the trial (e.g., active autoimmune disease or uncontrolled diabetes)
* No refractory nausea and vomiting, chronic gastrointestinal disease (e.g., inflammatory bowel disease), or significant bowel resection that preclude adequate absorption
* No psychiatric disorder precluding understanding of information on trial-related topics, giving informed consent, or interfering with adherence for oral drug intake
* No uncontrolled hypertension (systolic BP > 150 mm Hg and/or diastolic BP > 100 mm Hg, measured repeatedly at more than two visits despite adequate treatment with at least two different antihypertensive drugs)
* No clinically significant (i.e., active) cardiovascular disease, including any of the following:

  * Cerebrovascular accident/stroke or myocardial infarction within the past 6 months
  * Unstable angina
  * NYHA class III-IV congestive heart failure
  * Serious cardiac arrhythmia or AV-block > 1, requiring medication during the trial and which might interfere with regularity of the trial treatment, or not controlled by medication
* No known hypersensitivity to trial drugs or any other component of the trial drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 30 days since other prior experimental drugs or participation in another clinical trial
* No prior fulvestrant, AZD6244, MEK inhibitors, RAF inhibitors, or endocrine therapies other than aromatase inhibitors (e.g., anastrazole, letrozole, or exemestane) or tamoxifen
* No more than 1 line of aromatase inhibitors (steroidal and nonsteroidal aromatase inhibitors are considered two different lines)
* No concurrent full-dose anticoagulation therapy (e.g., low molecular weight heparin, acenocoumarol, phenprocoumon, or analogues)

  * Prophylactic doses of anticoagulation or antiplatelet may be allowed
* No concurrent radiotherapy
* No other concurrent anticancer therapy or experimental drugs
* Concurrent bisphosphonate allowed provided the investigator rules out tumor progression

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Disease control (sum of complete response, partial response, and stable disease) at 24 weeks or more according to RECIST 1.1 criteria | at 24 weeks or more according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Adverse events | according to NCI CTCAE v 4.0
Overall response | according to RECIST 1.1
Progression-free survival | will be calculated from randomization until documented tumor progression or death, whichever occurs first.
Time to treatment failure | will be calculated from randomization to discontinuation of all trial treatment due to any reason
Duration of response | will be calculated from the time that measurement criteria are met for the first time until documented tumor progression.
Overall survival | Overall survival will be calculated from registration until death

CONTACTS AND LOCATIONS:
Overall Officials: Khalil Zaman, MD, Study Chair — Centre Hospitalier Universitaire Vaudois; Lucien Perey, MD, Study Chair — Hopital de Morges; Patrick Neven, MD, PhD, Study Chair — University Hospital, Gasthuisberg
Locations (17):
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Gasthuisberg, Leuven
- Switzerland (15):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Graubuenden, Chur
  - Brustzentrum Thurgau at Kantonsspital Frauenfeld, Frauenfeld
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Luzern, Luzerne
  - Oncology Institute of Southern Switzerland - Mendrisio, Mendrisio
  - Hopital de Morges, Morges
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - City Hospital Triemli, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zaman K, Winterhalder R, Mamot C, Hasler-Strub U, Rochlitz C, Mueller A, Berset C, Wiliders H, Perey L, Rudolf CB, Hawle H, Rondeau S, Neven P. Fulvestrant with or without selumetinib, a MEK 1/2 inhibitor, in breast cancer progressing after aromatase inhibitor therapy: a multicentre randomised placebo-controlled double-blind phase II trial, SAKK 21/08. Eur J Cancer. 2015 Jul;51(10):1212-20. doi: 10.1016/j.ejca.2015.03.016. Epub 2015 Apr 16. PMID 25892646